CLINICAL TRIAL: NCT00035750
Title: Risk Factors for Atherogenesis in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1054; R01HL062897 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus, Insulin-dependent; Heart Diseases; Diabetes Mellitus
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Diabetes Mellitus, Type 1; Heart Diseases; Diabetes Mellitus

SUMMARY:
To determine risk factors for atherogenesis in Type 1 diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

Individuals with Type 1 diabetes have substantially higher risk for premature atherosclerotic vascular disease (ASVD) than the general population. Risk factors for the development of ASVD have been identified, but linking them to initiation of atherosclerosis was not feasible until recently. Advances in non-invasive imaging now permit early detection of changes in blood vessel function and structure. This imaging provides an opportunity to evaluate risk factors for ASVD and vascular status in a cohort at a critical time for development and early progression of ASVD.

DESIGN NARRATIVE:

Subjects were enrolled from 1987-1992 and were followed from diabetes diagnosis. Standardized protocols for examinations and interviews were implemented and the data base included a valuable longitudinal plasma bank. Because incident cases were enrolled, information was collected from diagnosis on children, adolescents and young adults currently without symptoms of atherosclerosis. The existing database was expanded, the existing resources were used including the plasma bank, and promising new and well established clinical research techniques were incorporated by: (i) measuring plasma lipid levels on stored plasma and on newly collected blood samples, (ii) measuring triglyceride levels on newly collected blood samples, (iii) measuring urinary albumin excretion rates on newly collected specimens (already measured from diagnosis to date), and (iv) assessing endothelial function by brachial artery ultrasound, (v) measuring the intima medial thickness (IMT) of the carotid artery by ultrasound, and (vi) measuring coronary calcium by computed tomography scanning. These activities allowed pursuit of the following specific aims: 1) to determine the relationship between established risk factors for atherosclerosis and the development of pre-clinical atherosclerosis, 2) to determine the relationship between endothelial dysfunction and carotid IMT, and 3) to determine the relationship between coronary artery calcification and carotid IMT. Such information was critical in directing further efforts toward primary prevention of atherosclerosis in individuals with Type 1 diabetes mellitus.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Mari Palta — University of Wisconsin, Madison

REFERENCES:
- [Background] Stein JH, Korcarz CE, Mays ME, Douglas PS, Palta M, Zhang H, Lecaire T, Paine D, Gustafson D, Fan L. A semiautomated ultrasound border detection program that facilitates clinical measurement of ultrasound carotid intima-media thickness. J Am Soc Echocardiogr. 2005 Mar;18(3):244-51. doi: 10.1016/j.echo.2004.12.002. PMID 15746714